CLINICAL TRIAL: NCT07379450
Title: Official Title: Effectiveness of Virtual Reality-enhanced Interventions on Preoperative Anxiety in Adults Undergoing Elective Surgery: A 3-arm Randomised Controlled Trial
Brief Title: Effectiveness of Virtual Reality-enhanced Interventions on Preoperative Anxiety in Adults Undergoing Elective Surgery
Acronym: VIPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sin Lun CHAN (Other)
Responsible Party: Sponsor-Investigator, Sin Lun CHAN, Principal Investigator, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIRB-2025-224-5
Record Dates: First submitted 2026-01-21; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Preoperative Anxiety
Keywords: Preoperative Anxiety; Virtual Reality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group 1 (Education approach) (Experimental): Participants in Virtual Reality Group 1 (Education approach) will receive a co-designed virtual reality educational 6-minute video via VR headset. The virtual reality educational video includes three main scenes, consisting of preoperative, intraoperative and postoperative content located at operating theatre reception, operating theatre, and post-anaesthetic care unit respectively.
  Interventions: Other: Virtual Reality
- Virtual Reality Group 2 (Distraction approach) (Experimental): Participants in Virtual Reality Group 2 (Distraction approach) will receive a virtual reality distraction 6-minute video via VR headset. The virtual reality distraction video includes immersive natural scenes with concurrent music, without educational component.
  Interventions: Other: Virtual Reality
- Control Group (No Intervention): Participants in control group will receive usual care only.

INTERVENTIONS:
Other: Virtual Reality — The Virtual Reality-enhanced Interventions on Preoperative Anxiety for adults undergoing elective surgery (VIPA) was developed based on theoretical basis, systematic review evidence, and qualitative study.
  Arms: Virtual Reality Group 1 (Education approach); Virtual Reality Group 2 (Distraction approach)

SUMMARY:
Brief Summary: Preoperative anxiety is a common phenomenon in surgical patients, with a pooled global prevalence of 48%. Surgical patients with preoperative anxiety may negatively impact their psychological health and surgical outcomes. Recent studies have revealed the promising effects of virtual reality-enhanced interventions to improve preoperative anxiety symptoms among adults undergoing elective surgery.

There is a lack of interventional studies to compare and evaluate the co-designed preoperative virtual reality-enhanced interventions in adult surgical patients.

This study aims to examine the effects of co-designed virtual reality educational video and virtual reality distraction video on preoperative anxiety symptoms, vital signs, Satisfaction with Life Scale (SWLS), and postoperative anxiety compared to usual care. This study will contribute by evaluating evidence-based, user-centered VIPA that may be effective for improving preoperative anxiety among adult surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Age aged ≥18 years old
* Surgical patients attending Nurse Pre-anaesthetic Assessment Clinic (NPAC)
* American Society of Anesthesiology (ASA) physical status ASA I or ASA II
* Able to communicate in Chinese

Exclusion Criteria:

* Patients who have a cognitive, communication or physical impairment precluding their ability to complete the study
* Patients who are prone to epilepsy or other neurological conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety | Baseline, Immediate post-intervention, Day of surgery
  Preoperative anxiety will be measured using the Short Chinese Version of the State-Trait Anxiety Inventory (Du et al., 2022). Items are rated on a 4-point Likert scale ranging from 1 to 4, with higher scores indicating higher anxiety. The Short Chinese Version of the State-Trait Anxiety Inventory demonstrates good psychometric properties.

SECONDARY OUTCOMES:
Heart rate | Baseline, Immediate post-intervention, Day of surgery
  Heart rate will be measured in beats per minute (bpm) using physiological monitors to provide a more objective measurement for anxiety.
Blood pressure | Baseline, Immediate post-intervention, Day of surgery
  Blood pressure will be measured in millimeters of mercury (mmHg) using physiological monitors to provide a more objective measurement for anxiety.
Temperature | Baseline, Immediate post-intervention, Day of surgery
  Temperature will be measured in degrees Celsius (°C) using tympanic thermometers to provide a more objective measurement for anxiety.
Life satisfaction | Baseline, Immediate post-intervention, Day of surgery, Post-operative day 7
  Life satisfaction will be measured using the Chinese version of Satisfaction with Life Scale (SWLS) (Diener et al., 1985). Items are rated on a 7-point Likert scale ranging from 1 to 7, with higher scores indicating higher life satisfaction. The Chinese version of Satisfaction with Life Scale (SWLS) demonstrates good psychometric properties (Wu & Yao, 2006).
Evaluation of Virtual reality-enhanced interventions questionnaire | Immediate post-intervention
  Virtual reality-enhanced interventions questionnaire was developed to evaluate virtual reality-enhanced interventions in terms of programme content, content adequacy, content usefulness, willingness to recommend others, satisfaction, and improvement suggestions. The questions are either 4-point Likert scale or open-end questions. The score ranges from 1 to 4, higher scores indicate higher satisfcation and higher agreement.
Postoperative anxiety | Post-operative day 7
  Postoperative anxiety will be measured using the Short Chinese Version of the State-Trait Anxiety Inventory (Du et al., 2022). Items are rated on a 4-point Likert scale ranging from 1 to 4, with higher scores indicating higher anxiety. The Short Chinese Version of the State-Trait Anxiety Inventory demonstrates good psychometric properties.

IPD SHARING:
Plan to Share IPD: No